CLINICAL TRIAL: NCT02386917
Title: Impact of Body Weight, Low Calorie Diet and Gastric Bypass on Drug Bioavailability, Cardiovascular Risk Factors and Metabolic Biomarkers
Brief Title: Impact of Body Weight and Weight Loss on Drug Bioavailability, Cardiovascular Risk Factors and Metabolic Biomarkers
Acronym: COCKTAIL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital of Vestfold (Other)
Collaborators: University of Oslo (Other); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Jøran Hjelmesæth, Professor, Head, The Hospital of Vestfold
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2013-2379
Record Dates: First submitted 2015-02-24; First posted 2015-03-12 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Gastric Bypass

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gastric bypass (Active Comparator): 40 patients will undergo gastric bypass
  Interventions: Procedure: Gastric bypass
- Very low calorie diet (Active Comparator): 40 patients will undergo a very low calorie diet
  Interventions: Behavioral: Very low calorie diet
- Gall bladder operation (No Intervention): 20 patients will be asked to undergo one pharmacokinetic study only, and then finish the study. They will not undergo any weight loss intervention.

INTERVENTIONS:
Procedure: Gastric bypass — Weight loss surgery
  Arms: Gastric bypass
Behavioral: Very low calorie diet — Non-surgical weight loss procedure
  Arms: Very low calorie diet

SUMMARY:
Drug bioavailability and disposition vary according to body weight and weight loss after bariatric surgery. This study evaluates the impact of body weight and weight loss on the pharmacokinetics of various probe drugs, and compares these effects in three groups of patients receiving either a gall bladder operation, gastric bypass or a very low calorie diet.

DETAILED DESCRIPTION:
This study aims to

1. to investigate the relationship between body composition and the liver/intestine activity and expression of proteins (drug metabolizing enzymes, transporters and regulatory factors) important for drug bioavailability and disposition in the range from normal to morbid obesity (the combined gastric bypass and cholecystectomy groups) at baseline.
2. to compare the short-term (6-week) and long-term (2 years) effect of gastric bypass (GBP) and a very low calorie diet (VLCD) (matched weight loss) on bioavailability and pharmacokinetics of probe drugs (caffeine, omeprazole, digoxin, midazolam, rosuvastatin, losartan) and biomarkers (and adjoining protein expressions) for cytochrome P450 (CYP)1A2, CYP2C9, CYP2C19, CYP3A, P-glycoprotein (gp) and organic anion-transporting polypeptide (OATP)1B1.
3. to compare the 3 study groups (GBP, VLCD and cholecystectomy) at baseline with respect to body composition, cardiovascular risk factors and metabolic biomarkers.
4. to compare the short-term (6-week) changes in glucose metabolism, blood pressure, blood lipids and body composition of matched weight loss and long-term effects (2 year) on body composition, cardiovascular risk factors and metabolic biomarkers, between the GBP and VLCD groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for GBP surgery or VLCD intervention for obesity as well as patients scheduled for cholecystectomy.
2. BMI ≥ 18.5 kg/m2
3. Able and willing to donate biopsies (as specified in the protocol) and for the GBP and VLCD patients also willing to perform follow-up 24 hour PK-investigations and other assessments as required by the clinical study protocol
4. Stable body weight (< 5 kg self reported weight change) during the last 3 months before inclusion.
5. Signed informed consent.

Exclusion Criteria:

* Concomitant treatment with drugs (according to available literature, appendix 3) and/or other factors that may influence the cocktail drug pharmacokinetics such as grapefruit juice, Seville oranges, Pomelo juice, St. Johns wort, tobacco and coffee/tea in close approximation to the investigations.
* Bradyarrhythmia, Wolff-Parkinson-White (WPW)-syndrome, atrioventricular block 2-3.
* Electrolyte disturbances (particularly hypokalemia or hypomagnesemia).
* Renal impairment: eGFR < 30 mL/min.
* Blood donations the last 4 months.
* Previous bariatric or upper gastrointestinal surgery.
* Diabetic patients treated with glitazones, insulin or sulfonylureas.
* Pregnancy (checked with HCG in urine at screening) and breast-feeding mothers.
* Known hypersensitivity (including allergy) to drugs included in the cocktail and/or local anesthesia.
* Anticoagulants with associated risk in combination with biopsies.
* Non-compliance with regards to visits and/or diet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-03-18 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Bioavailability of drugs (1) | 0 hours and 0.25, 0.5, 1, 1.5, 2, 3, 4, 4.25, 4.5, 5, 5.5, 6, 8, 10*, 12*, 23 and 24 hours following administration
  Changes in absolute bioavailability (Area Under Curve - oral / Area Under Curve -intravenous) of midazolam after Gastric Bypass and Very Low Calorie Diet, respectively.
Bioavailability of drugs (2) | 0 hours and 0.25, 0.5, 1, 1.5, 2, 3, 4, 4.25, 4.5, 5, 5.5, 6, 8, 10*, 12*, 23 and 24 hours following administration
  Changes in bioavailability (Area Under Curve - oral) of caffeine, losartan, digoxin, rosuvastatin and omeprazole after Gastric Bypass and Very Low Calorie Diet, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Jøran Hjelmesæth, Professor, Principal Investigator — The Hospital of Vestfold
Locations (1):
- HVestfold, Tønsberg, Vestfold, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karlsson C, Johnson LK, Greasley PJ, Retterstol K, Hedberg J, Hall M, Hawker N, Robertsen I, Havsol J, Hertel JK, Sandbu R, Skovlund E, Olsen T, Christensen H, Jansson-Lofmark R, Andersson S, Asberg A, Hjelmesaeth J. Gastric Bypass vs Diet and Cardiovascular Risk Factors: A Nonrandomized Controlled Trial. JAMA Surg. 2024 Sep 1;159(9):971-980. doi: 10.1001/jamasurg.2024.2162. PMID 38959017
- [Derived] Kvitne KE, Asberg A, Johnson LK, Wegler C, Hertel JK, Artursson P, Karlsson C, Andersson S, Sandbu R, Skovlund E, Christensen H, Jansson-Lofmark R, Hjelmesaeth J, Robertsen I. Impact of type 2 diabetes on in vivo activities and protein expressions of cytochrome P450 in patients with obesity. Clin Transl Sci. 2022 Nov;15(11):2685-2696. doi: 10.1111/cts.13394. Epub 2022 Sep 8. PMID 36037309
- [Derived] Eide Kvitne K, Hole K, Krogstad V, Wollmann BM, Wegler C, Johnson LK, Hertel JK, Artursson P, Karlsson C, Andersson S, Andersson TB, Sandbu R, Hjelmesaeth J, Skovlund E, Christensen H, Jansson-Lofmark R, Asberg A, Molden E, Robertsen I. Correlations between 4beta-hydroxycholesterol and hepatic and intestinal CYP3A4: protein expression, microsomal ex vivo activity, and in vivo activity in patients with a wide body weight range. Eur J Clin Pharmacol. 2022 Aug;78(8):1289-1299. doi: 10.1007/s00228-022-03336-9. Epub 2022 Jun 1. PMID 35648149
- [Derived] Hjelmesaeth J, Asberg A, Andersson S, Sandbu R, Robertsen I, Johnson LK, Angeles PC, Hertel JK, Skovlund E, Heijer M, Ek AL, Krogstad V, Karlsen TI, Christensen H, Andersson TB, Karlsson C. Impact of body weight, low energy diet and gastric bypass on drug bioavailability, cardiovascular risk factors and metabolic biomarkers: protocol for an open, non-randomised, three-armed single centre study (COCKTAIL). BMJ Open. 2018 May 29;8(5):e021878. doi: 10.1136/bmjopen-2018-021878. PMID 29844102